CLINICAL TRIAL: NCT06248034
Title: A Pilot Feasibility Study Comparing Smartphone Home-based Rehabilitation Program Against the Usual Hospital and Outpatient Physiotherapy Care on Clinical and Cost Effectiveness for Total Knee Replacement Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Rootally AI PTE LTD (Unknown)
Responsible Party: Principal Investigator, Eleanor Chew Shuxian, Senior Principal Physiotherapist, Singapore General Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/2482
Record Dates: First submitted 2024-01-17; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Knee Arthropathy
Keywords: Knee Arthroplasty;; Orthopedic Procedures;; Outcome Assessments;; Self- Help Devices;; Technology;; Knee: Treatment Outcome

STUDY DESIGN:
Intervention Model Description: The investigators will perform stratified randomization by surgeons, are evenly distributed between the 2 treatment arms. Arm 1: Smartphone Home-based Rehabilitation Program (N=15); Arm 2: Hospital-based rehabilitation program (N=15).
Who Masked: Outcomes Assessor
Masking Description: To reduce bias, the research assistant collecting assessment data will be blinded to treatment allocation. Participants will also be instructed not to reveal details about their group assignment to the outcome assessor to maintain blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants for Smartphone Home-based Rehabilitation Program (N=15) (Experimental): Study participants will be recruited from orthopaedic surgeons in Singapore General Hospital. Study participants will be recruited during their outpatient appointment session at the outpatient orthopaedic specialist clinic pre-admission clinic.
  Interventions: Device: Smartphone application with tele-monitoring rehabilitation
- Participants for Hospital-based rehabilitation program (N=15) (Experimental): Study participants will be recruited from orthopaedic surgeons in Singapore General Hospital. Study participants will be recruited during their outpatient appointment session at the outpatient orthopaedic specialist clinic pre-admission clinic.
  Interventions: Procedure: Hospital-based rehabilitation program

INTERVENTIONS:
Device: Smartphone application with tele-monitoring rehabilitation — This Smartphone application includes an automated criterion-based progression based on participant's regular recorded self-measurement of knee range-of-motion and five-repetition-sit-to-stand. The rehabilitation program is designed to (i) increase knee range-of-motion, (ii) strengthen lower limb strength, (iii) improve postural balance, and (iv) improve physical function.
  Arms: Participants for Smartphone Home-based Rehabilitation Program (N=15)
Procedure: Hospital-based rehabilitation program — Participants will be provided with the usual preoperative, inpatient physiotherapy and a physiotherapy house visit within the first 2-weeks postoperation. Participants will receive exercises, patient education, manual therapy and other modalities that were prescribed and progressed at the project physiotherapist's discretion.
  Arms: Participants for Hospital-based rehabilitation program (N=15)

SUMMARY:
Knee osteoarthritis (OA) is a common, chronic, and costly condition whilst total knee replacement (TKR) is a common orthopaedic surgical intervention. In Singapore, after TKR surgery, nearly all patients who are home discharged are referred to hospital-based outpatient rehabilitation. Although outpatient rehabilitation attendance is associated with better functional outcomes, access to rehabilitation care is limited as outpatient rehabilitation is costly and inconvenient for patients and their caregivers, resulting in suboptimal adherence.

A smartphone home-based rehabilitation program provides the best access to rehabilitation care and is a potential alternative for the majority of patients who do not require intensive "hands-on" rehabilitation therapy.

The primary aim of this randomized controlled trial is to compare patient functional outcomes and cost-effectiveness of this innovative smartphone home-based exercise program versus that of currently standard, hospital-based outpatient rehabilitation program among post TKR patients in the Department of Physiotherapy, Singapore General Hospital.

DETAILED DESCRIPTION:
Thirty patients undergoing TKR for knee OA will be randomly assigned to receive either smartphone home-based rehabilitation program or hospital-based rehabilitation program following surgery for a rehabilitation period of 24 weeks. The primary patient functional outcome will be fast gait speed. Outcomes will be assessed preoperatively, at 12-week and 24-week after surgery by an assessor masked to group allocation.

If shown to be non-inferior to the standard outpatient rehabilitation, smartphone home-based exercise program can be recommended as a cost effective treatment option for patients with TKR.

ELIGIBILITY:
Inclusion Criteria:

1. Primary unilateral total knee replacement
2. Age >= 45 years
3. Under the Enhanced Recovery After Surgery (ERAS) programme (discharge on post-operative day 0/1)
4. Able to ambulate independently without an assistive device
5. Willingness to be randomized to either smartphone home-based rehabilitation program or outpatient rehabilitation
6. Ability to provide informed consent
7. Able to operate phone application and use online platform
8. Able to read and understand English or Mandarin

Exclusion Criteria:

1. Rheumatoid arthritis and other systemic arthritis
2. Significant back or other non-knee pain
3. A previous history of stroke and other major neurological conditions
4. An intention to transfer to step-down care facilities post-operatively

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
Gait speed: | Pre-Operative, Week 12 & Week 24
  This provides a performance-based measure of physical function. As participants walk a 10-metre walkway at their usual and fast pace.

SECONDARY OUTCOMES:
Physical function: | Pre-Operative, Week 12 & Week 24
  The physical function will be measured using the subscale of Knee Osteoarthritis Outcome Score (KOOS) and Global Rating Scale, which are designed to evaluate the patient's opinion about their knee and associated problem.
Muscle strength: | Pre-Operative, Week 12 & Week 24
  One-repetition Maximum(1RM) is a measure of the maximal weight a participant can lift with one repetition.
Knee pain: | Pre-Operative, Week 12 & Week 24
  Knee pain intensity while navigating stairs, walking, standing and performing a sit-to-stand will be measured using the 10-point numeric pain rating scales (NPRS).
  0 - No pain 10 - Extremely painful
Knee range-of-motion: | Pre-Operative, Week 12 & Week 24
  A long-arm goniometer will be used to measure active-assisted knee flexion and extension range-of-motion with the participants in supine position.
Stair climb test: | Pre-Operative, Week 12 & Week 24
  This assesses the participants' ability to ascend and descend stairs, their lower limb strength, balance and endurance. The timing required for participants to ascend one flight of stairs, turn around and descend the same flight of stairs will be taken. The stair climb test is a measure that is performed as part of standard clinical practice.
5-repetition-sit-to-stand test: | Pre-Operative, Week 12 & Week 24
  A test to assess participants' ability to rise from a chair and return to the sitting position. The time taken for participant to stand up and sit down five times as fast as possible from standard chair (43-47cm) without the use of their hands will be recorded. This test is a measure that is performed as part of standard clinical practice and is also a measure of lower limb strength and dynamic balance.
30 seconds-sit-to-stand test: | Pre-Operative, Week 12 & Week 24
  A test to assess participants' ability to rise from a chair and return to the sitting position within 30seconds from standard chair (43-47cm) without the use of their hands will be recorded.

OTHER OUTCOMES:
Quality of the mobile application: | Week 12 & Week 24
  The Mobile Application Rating Scale:user version (uMARS) will be used to measure the quality of the application. This scale assesses the engagement, functionality, and aesthetics of the application.
  1- Strongly disagree 5- Strongly agree
Treatment credibility: | Week 24
  Treatment credibility will be measured using the treatment credibility scale. Participants will rate their confidence about the benefits of the intervention on a 11-point Likert scale, with 0 indicating "not confident" and 10 indicating "extremely confident".
Perceived usefulness and ease of use: | Week 12 & Week 24
  These measures will be measured on a 10-point numeric scale. 0 - Not at all satisfied 10-Extremely satisfied
Participants satisfaction: | Week 12 & Week 24
  Immediately post intervention at 12-week and at 24-week time-point, participants will rate their satisfaction with rehabilitation on a 20-cm visual analogue scale, with 0 cm indicating "no satisfaction" and 20 cm indicating "complete satisfaction".
EQ5D-5L: | Week 12 & Week 24
  The EQ5D-5L is a standardised instrument to measure health related quality of life in cost-effectiveness analysis.
Adverse effects: | Week 24
  The adverse effects for participants randomized to the hospital-based rehabilitation group would be, such as falls or reports of injuries during the exercises, they will be monitored by questioning participants at each outpatient visit by the treating physiotherapists.
  For participants randomized to the smartphone home-based group, weekly exercise outcome reports will be sent to a research coordinator. Based on regular reports of participant's knee range-of-motion, 5-repetition-sit-to-stand, ability to perform exercises and activities, the physiotherapist will provide hospital-based rehabilitation to participants who are deemed to have deviated from the expected course of recovery and are at risk for poor functional outcomes.
Implementation outcomes: | Week 12 & Week 24
  The feasibility and acceptability of implementing the smartphone home exercise program will be evaluated. Specifically, the investigators will compute the proportion of eligible patients and evaluate the reasons for non-participation. Study participants will be asked to indicate, prior to surgery, their preference for the mode of treatment (smartphone home-based exercise program or hospital-based rehabilitation). Immediately post intervention at the 24-week time-point, participants will rate their satisfaction with home exercise program.

IPD SHARING:
Plan to Share IPD: No